CLINICAL TRIAL: NCT06794814
Title: Oral Function Improvement Through Oral Exercise: Gender Differences in Community-Dwelling Older Adults
Brief Title: Program of Community Oral Function Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NYCU113040AF
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Oral Hypofunction
Keywords: Oral exercises, community-dwelling elderly, oral function, prevention of chewing and swallowing disorders
MeSH Terms: conditions — Deglutition Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental)
  Interventions: Behavioral: oral exercise

INTERVENTIONS:
Behavioral: oral exercise — The oral exercise protocol included several physical components, namely neck and shoulder stretching, cheek puffing exercises, tongue exercises, salivary gland massage, and oral diadochokinesis.

SUMMARY:
The purpose of this study examined the effects of oral exercise on oral function among older adults in Taiwan, focusing on gender-related outcome differences.

Seventy-seven community-dwelling older adults aged 65 and above participated in a six-week oral exercise program, performed before each meal.

After six-week, the participants were examed the salivary secretion, swallowing ability (RSST), oral diadochokinesis, bite force, quality of life (assessed by OHIP-14) and EAT-10.

DETAILED DESCRIPTION:
Objective: Elderly individuals with systemic diseases and disabilities face an elevated mortality risk, with oral functional decline further contributing to both oral and systemic health challenges. Given the rising prevalence of reduced oral function in older adults, this study aims to evaluate the effectiveness of oral exercise training on improving oral function and preventing functional decline. Additionally, the study examines potential gender differences in response to the intervention.

Methods: Seventy-seven community-dwelling older adults aged 65 and above participated in a six-week oral exercise program, performed before each meal. The study measured changes in oral function post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 65

Exclusion Criteria:

* incomplete data
* failed to perform the assigned daily exercise
* unable to adhere to the protocol and steps outline in the oral exercise video

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Oral Function Improvement Through Oral Exercise: Gender Differences in Community-Dwelling Older Adults | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lun Hsu, Distinguished professor, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No